CLINICAL TRIAL: NCT03437993
Title: Recollect the Game: A Novel Treatment for Executive Functioning Deficits in Adults With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Recollect_ADHD
Record Dates: First submitted 2018-02-07; First posted 2018-02-19 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Adult ADHD
Keywords: ADHD; executive functioning; game
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recollect (Experimental): Recollect is a video game which incorporates scientifically supported renditions of N-Back, Item Span, and Multiple-Identity tracking tasks. These tasks are independently shown to improve working memory in a manner that transfers to untrained tasks.
  Interventions: Other: Recollect, the game
- Tetris (Sham Comparator): Tetris is a video game which has not been shown to have any benefits in the improvement of executive functioning.
  Interventions: Other: Tetris

INTERVENTIONS:
Other: Recollect, the game — "Recollect" is a working memory training game
  Arms: Recollect
Other: Tetris — App-based video game where shapes are rotated and placed to fit a grid
  Arms: Tetris

SUMMARY:
Adults who have attention deficit hyperactivity disorder (ADHD) suffer from significant occupational, academic and social problems, many of which are believed to be a result of problems with executive functioning. Executive functioning refers to a group of neuro-psychological functions which include sustained attention, working memory, verbal fluency, as well as motor and mental processing speed. Individuals with ADHD have been shown to have deficits in executive functioning independent of IQ, co-occurring psychiatric disorders, gender, and ADHD subtype. "Recollect" is an application (App) based working memory training video game where participants conduct 3-different adaptive working memory tasks. In each of these tasks participants are presented with a set of stimuli to be remembered while playing a simple platform game where they help navigate an astronaut across the screen and dodge obstacles. Recollect has been designed for all age groups to an interesting, fun and effective brain-training activity. The memory tasks included in the game have been independently shown to improve working memory in a manner that transfers to untrained tasks.

The purpose of this study is to evaluate the effects of playing Recollect versus Tetris for 20 minutes per day, 5 days per week over a 4 week period, on executive functioning deficits in individuals who have Adult ADHD.

DETAILED DESCRIPTION:
The primary objective is to evaluate the effects of playing Recollect versus Tetris for 20 minutes per day, 5 days per week over a 4 week period, on executive functioning deficits in individuals who have Adult Attention Deficit Hyperactivity Disorder (ADHD).Consenting participants will be screened using the Mini International Neuropsychiatric Interview for DSM-5 (MINI) to confirm ADHD diagnosis. Participants will be asked to download either Recollect or Tetris on their own mobile device. Following a training/orientation session, they will be asked to spend 20 minutes per day at least 5 days per week playing Recollect or Tetris over a 4 week period. At Week 4, study staff will check the time log on the Recollect/Tetris App to confirm how much time was spent playing the game. Participants will be asked to complete two ADHD symptom severity scales, as well as App-based neurocognitive testing at baseline (Week 0) and endpoint (Week 4).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 and older who own a mobile device such as a Smartphone or tablet.
2. Current diagnosis of Adult ADHD, at any stage of treatment.
3. Comorbid psychiatric conditions will be allowed.
4. Medication or psychotherapy must have been stable (no dose changes) for 4 weeks prior to study participation.
5. Must be able to read, write and understand English.

Exclusion Criteria:

1. Participant does not own a Smartphone or tablet.
2. No dose changes during the 4 week study period.
3. No initiation of new psychological therapy or counselling during the 4 week study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on The Behavioral Rating Inventory of Executive Functioning - Adult Version (BRIEF-A) | Change from baseline to week 4
  It is a validated, clinician-rated scale, measuring executive functioning. The scale includes 75 items that rates patient symptoms on a 3-point Likert scale (1 = behavior is never observed to 3 = behavior is often observed). Scores range from 75 to 225: Higher scores indicate greater impairment in executive functioning.

SECONDARY OUTCOMES:
Change from baseline on the Barkley Adult ADHD Rating Scale (BAARS-IV) | Change from baseline to week 4
  Self-report scale evaluating ADHD symptoms. Symptom count scores range from 1 to 27, with higher scores indicating more ADHD symptoms. Total scores range from 27 to 108, with higher scores indicating greater severity of symptoms.
Change from baseline on an App-based neuro-cognitive battery | Change from baseline to week 4
  A number of neuro-cognitive executive functioning tests, which will be administered via a smartphone application

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided